CLINICAL TRIAL: NCT07173296
Title: The Effect of Single and Multiple Application of In-office Dental Bleaching on Tooth Sensitivity and Bleaching Efficacy: a Single-blind Randomized Controlled Trial
Brief Title: The Effect of Bleaching Application Mode on Bleaching-induced Tooth Sensitivity.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah University Hospital (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Ghada Maghaireh, Principal Investigator, King Abdullah University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0541-2024
Record Dates: First submitted 2025-08-27; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Tooth Sensitivity
Keywords: Sensitivity; Application mode; in-office bleaching
MeSH Terms: conditions — Dentin Sensitivity; Hypersensitivity | interventions — pola office

STUDY DESIGN:
Intervention Model Description: This study will be a randomized, single-blind (evaluators), split-mouth with an equal allocation rate between groups. Blocked randomization will be performed (block size of 2) to guarantee equal-sized groups with an equal allocation ratio at www.sealedenvelope.com. A third party not involved in the study will prepare consecutively numbered, opaque, and sealed envelopes containing information identifying the groups. The group that will be identified in the envelope will be corresponded to the treatment that will be performed on the right upper hemiarch, and the left hemiarch will receive the alternate treatment.
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opalescence (Experimental): Group 1: Opalescence XTra Boost 40% HP (OB) [Ultradent, Salt Lake, UT, USA] which will be used in a split-mouth design for a single application for 40 minutes and 2 applications for 20 minutes each.
  Interventions: Other: Opalescence XTra Boost 40% HP
- PolaOffice (Experimental): Group 2: Pola Office Plus 37.5% HP (PO) [SDI, Bayswater, Australia] which will be applied in a split-mouth design for a single 32 minutes and 4 applications of 8 min each
  Interventions: Other: Pola Office Plus 37.5% HP

INTERVENTIONS:
Other: Opalescence XTra Boost 40% HP — In-office tooth bleaching material
  Arms: Opalescence
Other: Pola Office Plus 37.5% HP — In-office tooth bleaching material
  Arms: PolaOffice

SUMMARY:
The aim of this study is to evaluate the effect of single versus multiple application protocols for in-office dental bleaching using two different bleaching gels (Pola Office Plus, SDI, 37.5% HP and Opalescence Boost, Ultradent, 40% HP) on the risk and intensity of tooth sensitivity, as well as the effect of the application protocol on the bleaching efficacy.

Null hypothesis: There is no difference in intensity and risk of tooth sensitivity between single and multiple application of each gel and the application protocol dose not present significant effect on the bleaching efficacy.

DETAILED DESCRIPTION:
IV. Materials and Methods:

The study will be conducted in the post graduated Restorative dentistry clinics at Jordan University of science and technology. Ethical approval will be obtained from the JUST institutional ethics and human research board (IRB) committee. All the participants will be examined in a dental chair after dental prophylaxis with pumice and water to check whether they meet the study's eligibility criteria (Table 1).

Sample size estimation:

The primary outcome of this study is the absolute risk of tooth sensitivity. The absolute risk of tooth sensitivity was reported to be approximately 90% (21,22) for the in-office bleaching. Thus, a minimum sample size of 30 patients will be required in each group to have an 80% chance of detecting (with an alpha of 5%) a decrease in the primary outcome measure from 90% in the multiple application protocol to 45% in the single application group.

Experimental design:

This study will be a randomized, single-blind (evaluators), split-mouth with an equal allocation rate between groups. Blocked randomization will be performed (block size of 2) to guarantee equal-sized groups with an equal allocation ratio at www.sealedenvelope.com. A third party not involved in the study will prepare consecutively numbered, opaque, and sealed envelopes containing information identifying the groups. The group that will be identified in the envelope will be corresponded to the treatment that will be performed on the right upper hemiarch, and the left hemiarch will receive the alternate treatment. The groups of the study are: Group 1: Opalescence XTra Boost 40% HP (OB) [Ultradent, Salt Lake, UT, USA] which will be used in a split-mouth design for a single application for 40 minutes and 2 applications for 20 minutes each. Group 2: Pola Office Plus 37.5% HP (PO) [SDI, Bayswater, Australia] which will be applied in a split-mouth design for a single 32 minutes and 4 applications of 8 min each. For the multiple application technique, the exact manufacturer's recommendation will be followed. For the single application technique, the sum of application time will be calculated for each product. Details regarding the bleaching agents and application protocols are provided in Table 2.

Study Intervention:

A lip and cheek retractor will be placed. The gingival tissues from the right first molar to the left first molar will be isolated using a light-cured resin dam to prevent the whitening gel from coming into contact with the gingival tissue. Participants' lips will be painted with Vaseline, and protective eyewear will be used. To aid in the isolation process, a plastic suction tip with high suction power will be used.

In Group 1, Opalescence XTra Boost 40% HP will be applied in a single 40-minute application or in two 20-minute applications in all maxillary incisors, canines, and premolars of the same patient. In Group 2, Pola Office Plus 37.5% HP will be applied in a split-mouth design for a single 32 minutes and 4 applications of 8 minutes in all maxillary incisors, canines, and premolars of the same patient.

After seven days, this procedure will be repeated using the same protocol. All participants will be instructed to brush their teeth using a supplied dentifrice (Colgate toothpaste maximum cavity protection 100 mL, Colgate-Palmolive Arabia, Dammam, Saudi Arabia).

Sensitivity evaluation:

Patient pain perception will be used to assess post-bleaching sensitivity using a 0-10 visual analog scale (VAS) and the Numerical Rating Scale (NRS) after each bleaching session in four different assessment periods: during treatment and up to 1 hour after bleaching, from 1 hour to 24 hours after bleaching, from 24 hours to 48 hours after bleaching and after 14 days of bleaching.

The VAS is a horizontal line with ten digits on it, ranging from 0 to 10, where 0 denotes no pain and 10 represents the worst possible suffering. The participants will be asked to identify their level of pain by marking the corresponding number. The NRS scale comprises scores to denote the intensity of pain (0 = none, 1 = mild, 2 = moderate, 3 = considerable, and 4 = intense). The stimulus-heat, cold, or another-that triggered sensitivity will be noted by the participants. For the 14-day follow-up period, the length of pain-whether it lasts for seconds, minutes, or hours-will be noted. In the multiple application protocol, the worst scores or numerical values obtained will be considered for statistical purposes. The values were organized into two categories: percentage of patients who reported tooth sensitivity at some time of treatment (absolute risk of sensitivity) and intensity of pain. The intensity results will be classified using the following scale for descriptive analysis purposes: 0 = none, 1-3 = mild, 4-6 = moderate, and 7-10 = severe.

Shade evaluation:

Shade will be recorded before the bleaching procedure, seven days later, and 30 days after the end of the bleaching treatment. The tooth shade will be evaluated subjectively using the VITA classical shade guide and Vita Bleached guide. A VITA easy shade spectrophotometer (VITA Easyshade V; VITA Zahnfabrik, Bad Säckingen, Germany) will also be used to objectively examine the shade of teeth. It is necessary to thoroughly hydrate the tooth before examining its color. For both devices, color will be checked at the middle third of the canine. The participants' tooth shades will be noted by a single assessor at baseline (before to whitening), immediately following bleaching, and at the three, seven, and fourteen-day follow-up intervals. To record the outcomes, digital cameras will be used to take pictures just after the whitening and at each shade assessment.

For the objective shade evaluation, an impression of the maxillary arch with high-putty silicon paste (Clonage, Nova DFL, Rio de Janeiro, RJ, Brazil) will be taken, and a window on the labial surface of the silicon guide will be created using a metal device with a 6-mm radius. The purpose of this is to standardize the area for color evaluation in all recall periods with the spectrophotometer. Color will be determined using the parameters of the digital spectrophotometer on which the following values will be indicated: L*, a*, and b*, where L* represented luminosity (the value from 0 [black] to 100 [white]), and a* and b* represented color along the red-green axis and the color along the yellow-blue axis, respectively. The difference between the baseline and each recall period (DE*) will be calculated using the following formula: DE* = [(DL*)2 þ (Da*)2 þ (Db*)2] 1/2. For the subjective evaluation, the 16 tabs of the shade guide (VITA classical, Vita Lumin, Vita Zahnfabrik, Bad Sa¨ckingen, Germany) and the 29 tabs of the shade guide (Vita Bleachedguide, Vita Lumin, Vita Zahnfabrik, Bad Sa¨ckingen, Germany) will be arranged from whitest to darkest.

ELIGIBILITY:
Inclusion Criteria:

* At least eight maxillary anterior teeth present.
* Age over 18
* The selected teeth have a mean shade of C2 or darker.
* Good general and oral health. (no visible plaque or gingivitis)
* No restorations or carious lesions on the buccal surfaces of the anterior teeth to be whitened
* No history of tooth sensitivity
* No use of a desensitizing agent or desensitizing toothpaste in the past six months
* No use of pain killer for the last 48 hours

Exclusion Criteria:

* Active caries and/or periodontal diseases (gingivitis and recession) or wasting diseases
* Smokers
* Pregnant/lactating women.
* Patients who have bleached their teeth previously.
* No schedule availability

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Tooth Sensitivity | Assess sensitivity during the bleaching, 1 hour after bleaching, 1 day, 2 days and 7 days after bleaching.
  Assessing reported tooth sensitivity by two scales.The VAS is a horizontal line with ten digits on it, ranging from 0 to 10, where 0 denotes no pain and 10 represents the worst possible suffering. The participants will be asked to identify their level of pain by marking the corresponding number. The NRS scale comprises scores to denote the intensity of pain (0 = none, 1 = mild, 2 = moderate, 3 = considerable, and 4 = intense).

SECONDARY OUTCOMES:
Change in teeth color | Shade will be recorded at base line before the bleaching procedure, seven days later, and 30 days after the end of the bleaching treatment.
  Assessing the change in tooth color by two ways. Subjectively using the VITA classical shade guide and Vita Bleached guide and objectively using the VITA easy shade spectrophotometer.

CONTACTS AND LOCATIONS:
Overall Officials: Ghada A Maghaireh, Principal Investigator — Jordan University of Science and Technology
Locations (1):
- Jordan University of Science and Technology, Irbid, Jordan

IPD SHARING:
Plan to Share IPD: No